CLINICAL TRIAL: NCT06773364
Title: An Investigator Initiated and Conducted, Prospective, Multicentre, Randomised Outcome-blinded Study of Pre-hospital Initiated Levetiracetam and Headposition in Patients With Presumed Acute Stroke
Brief Title: Early Initiated Ambulance-delivered Levetiracetam and Headposition in Hyper-acute Stroke Trial
Acronym: EAST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-228
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-01

CONDITIONS: Suspected Stroke
Keywords: Ambulance; Acute stroke; Levetiracetam; Head position; intervention
MeSH Terms: conditions — Stroke | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Levetiracetam (Experimental): Prophylactic use of LEV in the ambulance
  Interventions: Drug: Levetiracetam
- Guide-recommended management (Active Comparator): Guide-recommended management
  Interventions: Other: Guide-recommended management
- Lie flat (Experimental): Lie flat
  Interventions: Other: The lying flat (0°) head position
- Sit up (Active Comparator): Sit up
  Interventions: Other: The sitting-up (≥30°) head position

INTERVENTIONS:
Drug: Levetiracetam — Intervention group - to commence IV levetiracetam 500mg as a single bolus in the ambulance, and then to continue as levetiracetam 500mg bid orally after admission to hospital in those with confirmed acute stroke for the next 14 days (at least 7 days if either dead or discharged from hospital if earlier). They will also receive standard management of acute stroke, whether the final diagnosis is ischaemic or ICH
  Arms: Levetiracetam
Other: Guide-recommended management — To receive stroke management according to standard local guidelines, but to avoid prophylactic use of an anti-seizure drug.
  Arms: Guide-recommended management
Other: The lying flat (0°) head position — Lie flat (0°) - in the ambulance as soon as possible until arrival at hospital.
  Arms: Lie flat
Other: The sitting-up (≥30°) head position — Sit up(30-60°) - in the ambulance as soon as possible until arrival at hospital.
  Arms: Sit up

SUMMARY:
This is an investigator initiated and conducted, multicentre, ambulance-delivered, prospective, randomised, open-label, blinded outcome (PROBE) study. EAST aims to evaluate the effects of pre-hospital levetiracetam and different head positions initiated in ambulance settings on the functional outcome of participants assessed at 90 days.

DETAILED DESCRIPTION:
EAST is a multicenter, ambulance-delivered, prospective, randomized controlled, open label blinded outcome assessment (PROBE) study to be conducted through a regional-cluster hospital network of investigators. A total of 2323 patients with suspected acute stroke will be recruited from approximately 50 hospitals in China. Potentially eligible patients will be recruited into the study by either of two mechanisms: (1) waver of consent to the intervention, and consent to follow-up obtained in hospital; or (ii) consent to the intervention through a brief written consent which is combined with a usual care consent form delivered in hospital for follow-up (if a waver of consent is not approved by the ethics committee). All patients will enter Part A and Part B at the same time, randomised allocation of intervention will be done in a 1:1 ratio in each part, using a central, automated, mobile phone Wechat mini program-based electronic randomization software according to minimization method stratified by ambulance systems, age (≥65 vs <65) and FAST(>2 vs =2). The intervention of Part A is to commence IV levetiracetam(LEV) 500mg as a single bolus in the ambulance and then to continue as LEV 500mg Bid orally after hospital admission for 14 days(at least 7 days if discharged or death early), compared to avoid prophylactic use of antiseizure drugs. Part B is to lie flat or sit up in the ambulance as soon as possible until hospital arrival. Ambulance staff will be well trained across the whole study to master mobile randomisation and simple key data collection. All information in ambulance, including basic demographics, randomised allocation, BP measurement and treatment details, will be collected through mobile phone based electronic database system connected with investigator clinicians in hospitals. Other relevant documents such as consent paper, BP chart will be handed over to hospital investigators. Endpoint assessment will be blinded to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years);
* Acute condition that is presumed due to acute stroke, defined on the FAST (Face, Arm, Speech, Time) screen (score ≥2 with an arm deficit);
* Time ≤2 hours from last seen well;
* Able to provide brief consent (if a waver of consent not approved by ethics committee).

Exclusion Criteria:

* coma (no response to painful stimulation);
* severe co-morbid disease (e.g. cancer, chronic airflow disease, severe dementia, severe heart failure, pre-existing disability [needing help with everyday activities]);
* history of epilepsy or seizure at onset;
* recent head injury;
* hypoglycaemia (glucose <2.8mmol/L);
* clear indications or contraindications (allergies) for levetiracetam;
* lactating women;
* clear indications for a particular head position or situations where either head position cannot be maintained (such as severe vomiting and inability to lie down, severe obesity with fatigue and difficulty sitting up, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2423 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional shift (improvement) in 7-level mRS scores | 90 days

SECONDARY OUTCOMES:
neurological severity on the National Institute of Health stroke scale (NIHSS) | 24 hours from randomization
  0-42, higher scores indicates worse severity
neurological severity on the National Institute of Health stroke scale (NIHSS) | 7 days
  0-42, higher scores indicates worse severity
health related quality of life on the EQ-5D-5L | 90 days
severe disability (mRS 3-5) | 90 days
death and/or severe disability (mRS 3-6) | 90 days
utility-weighted-mRS (UW-mRS) | 90 days
proportion of hospital discharge at Day 7 | 7 days
living circumstances questions | 90 days
  living at home [the individual's own or that of a family member] or living at an institution(hospital, care facility, or other)
any seizures during follow-up | 90 days, 6 months, 12 months
  assessed by 6 screening questions modified from the Canadian Longitudinal Study on Aging-Epilepsy Algorithm (CLSA-EA)
haematoma volume | at hospital admission and 24 hours
  in patients with final diagnosis of ICH
Hematoma expansion | 24 hours
  in patients with final diagnosis of ICH

CONTACTS AND LOCATIONS:
Overall Officials: Gang Li, PhD, MD, Principal Investigator — Tongji University, School of Medicine, Shanghai East Hospital; Craig Anderson, MD, PhD, Principal Investigator — Fudan University; Lili Song, PhD, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Si County People's Hospital, Suzhou, Anhui
  - Shanghai East Hospital, Shanghai, Shanghai Municipality